CLINICAL TRIAL: NCT05348395
Title: Mechanism of Monocyte Priming in Humans - a Feeding Trial
Brief Title: Monocyte Priming When Consuming a Western Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00083476; R01HL153120 (NIH)
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-12

CONDITIONS: Heart Diseases
Keywords: heart disease; Western Diet; high-calorie diet
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental diet (Experimental): The experimental diet will provide 15% of calories from saturated fat and 14% of calories from fructose with a goal of providing 1.25x total energy needs
  Interventions: Other: Experimental diet

INTERVENTIONS:
Other: Experimental diet — Participants that successfully complete the run-in phase will participate in the experimental diet for 8 weeks of feeding. The Participants' adherence will be monitored using direct observation, written daily food diaries, and food waste inventory (i.e., participants are trained to estimate portion of uneaten foods). Participants will be asked to eat one meal onsite 2-3 weekdays (e.g., Monday, Wednesday, and Friday), at which time they will receive meals and snacks for the remainder of that day and enough until the next scheduled visit.

SUMMARY:
To determine the mechanism of monocyte priming in humans, the study team will conduct a complete feeding trial in normal weight and metabolically healthy human subjects (20-45 years of age) using a western diet (WD), characterized as being high-saturated fat, high-fructose, and high-calorie for 8 weeks.

DETAILED DESCRIPTION:
The goal is to challenge metabolically healthy human subjects with a high-calorie, Western diet for 8 weeks to identify the metabolite(s) responsible for monocyte priming and use redox proteomics, RNAseq and Chipseq to determine the genes and pathways involved in monocyte priming in humans. To reflect some key components of the typical Western intake, the Study Team will compose the diet to be high in saturated fat (15% of total energy intake) and fructose (14% of total energy intake) with excess energy intake that is 25% higher than estimated total energy expenditure. A total of 30 participants, including 15 men and 15 women, will complete a run-in phase where weight stability will be achieved on the control diet. After weight is stabilized during the run-in period, participants will enter the experimental phase of the dietary intervention, where overfeeding will begin with additional calories provided by the key nutrients as noted above. Participants will be monitored throughout the feeding trial. After completion of the 8-week overfeeding period, individuals will be allowed to return to a normal dietary intake. All study participants will be given access to counseling for weight reduction should it be needed following the overfeeding period.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-45
* Planning to be available for the entire study period
* Able to speak and read English
* Normal weight (body mass index 18.5-24.9 kg/m2)
* Able to eat the prescribed diet
* Non-smoker

Exclusion Criteria:

* Excessive alcohol consumption
* History of chronic cardiometabolic disease or major risk factor, including diabetes, hypertension, hyperlipidemia, heart disease
* History of prior surgical procedure for weight control or liposuction
* Use of weight loss medications in previous 6 months
* Recent self-reported weight change
* Severe pulmonary disease requiring supplemental oxygen
* Abnormal renal or liver function
* History of non-skin cancer in the past 5 years
* Regular use of medications (prescribed or over-the-counter) that affect blood pressure, lipids, glucose, inflammation, or body weight
* Works night shifts
* Exercise per week > 420 minutes total for moderate activity or > 210 minutes for vigorous activity
* Any medical or behavioral indication that would make participation unsafe based on the judgement of the study physician
* Pregnant or lactating women
* Known or discovered intolerances, allergies or difficulty consuming any of the foods included in the study diets

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Measurement of Mitogen-activated protein kinase phosphate 1 (MKP-1) activity | change in at the endpoint of week 8
  Analyze plasma from all subjects for their plasma lipid composition using an unbiased lipidomics approach in order to identify the lipid species responsible for monocyte priming

SECONDARY OUTCOMES:
Measurement of Monocyte protein S-glutathionylation | change in at the endpoint of week 8
  To identify which proteins alter their S-glutathionylation status (and possibly their expression levels) in response to HCD-induced monocyte priming, and which signaling pathways are altered in these cells.
  Isolate S-glutathionylated proteins from all samples and subject them to redox proteomics approach to identify S-glutathionylated proteins and to determine the extent and directionality of modifications on their cysteine residues.

OTHER OUTCOMES:
Ribonucleic acid (RNA) analysis | change in at the endpoint of week 8
  Determine the genes and pathways involved in monocyte priming in humans. Quantify mRNA expression of all transcripts in expressed monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Jamy Ard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Our plan to share materials and manage intellectual property will adhere to the NIH Grant Policy on Sharing of Unique Research Resources including the Sharing of Biomedical Research Resources.
Supporting Information: Study Protocol, CSR
Time Frame: before or immediately after publication
Access Criteria: upon request

DOCUMENTS (1):
  • Informed Consent Form (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT05348395/ICF_000.pdf